CLINICAL TRIAL: NCT01017211
Title: Does Auricular Acupuncture Improve Tolerance to Electromyography (EMG) Testing?
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Trevor A. Dyson-Hudson, M.D., Kessler Foundation Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-654-09
Record Dates: First submitted 2009-11-18; First posted 2009-11-20 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Pain
Keywords: Pain; Electromyography; Acupuncture; Randomized controlled trial; Rehabilitation
MeSH Terms: conditions — Pain | interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- auricular acupuncture protocol (Experimental)
  Interventions: Other: auricular acupuncture
- sham auricular acupuncture (Sham Comparator)
  Interventions: Other: auricular acupuncture

INTERVENTIONS:
Other: auricular acupuncture — Experimental group to receive ear needles in the Battlefield Acupuncture points.
  Sham group to receive ear needles at points thought to be ineffective but standardized.

SUMMARY:
Needle Electromyography (EMG) is an important test used to assess muscle and nerve function, but the test can be uncomfortable. It is currently not standard practice to provide any pain-relieving intervention for this procedure. The purpose of this research study is to determine whether auricular (ear) acupuncture will make EMG testing less painful.

ELIGIBILITY:
Inclusion Criteria:

* Gender: male or female
* Of any racial or ethnic group
* Adult between the ages 18 to 65 years
* Healthy
* Normal sensation and strength
* Pain approximately the same on each side of body with no major difference between right and left sides
* Can understand and are able to complete the outcomes questionnaires which will be explained before the study protocol begins

Exclusion Criteria:

* Pregnant or actively trying to become pregnant
* Diabetes mellitus or other systemic disease which may affect nerve function
* History of a neurologic disorder or other cause for abnormal sensation or weakness
* Have had recent trauma to an upper arm, hand or ear
* Have scars or burns on an upper arm, hand or ear that causes abnormal or decreased sensation
* Taking pain medications on a regular basis
* Have a bleeding or clotting disorder
* Taking blood thinners, such as aspirin, heparin, enoxaparin (Lovenox), clopidogrel (Plavix) or coumadin (Warfarin)
* Have received chemotherapy or radiation
* Have a permanent pacemaker
* Have a serious psychiatric disorder (such as schizophrenia)
* More sensitive to pain on one side of my body more than the other

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | pre- and post- intervention

SECONDARY OUTCOMES:
Global Impression of Change | pre- and post- intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Cole, M.D., Study Director — Kessler Institute for Rehabilitation
Locations (1):
- Kessler Institute for Rehabilitation, West Orange, New Jersey, United States